CLINICAL TRIAL: NCT05210101
Title: A Safety and Tolerability Study of Sotrovimab (VIR-7831) Prophylaxis Against COVID-19 Infection in Immunocompromised Individuals With Impaired SARS-CoV-2 Humoral Immunity
Brief Title: A Safety and Tolerability Study of Sotrovimab (VIR-7831) Prophylaxis Against COVID-19 in Immunocompromised Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sophia Koo, M.D. (Other)
Collaborators: Massachusetts General Hospital (Other); Dana-Farber Cancer Institute (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Sophia Koo, M.D., Sponsor-Investigator, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-755
Record Dates: First submitted 2022-01-25; First posted 2022-01-27 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: SARS CoV 2 Infection
Keywords: Prophylaxis; Immunocompromised host; Transplant; Monoclonal antibodies
MeSH Terms: conditions — COVID-19 | interventions — sotrovimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sotrovimab (Other): Two intravenous (IV) doses of sotrovimab were be administered in total - the first on Treatment Day 1 (500mg) and the second on Treatment Day 2, approximately 8-14 weeks after the first dose, at a higher 2000mg dose, in light of the reduced antiviral susceptibility of the BA.2 subvariant to sotrovimab, with the dosing interval determined by theoretical modeling of the duration of efficacy of sotrovimab as antiviral prophylaxis based on the rising prevalence of the Omicron BA.2 subvariant.
  Interventions: Drug: Sotrovimab

INTERVENTIONS:
Drug: Sotrovimab — Two intravenous (IV) doses of sotrovimab were administered over the study period, the first 500mg, and the second 2000mg, in light of the reduced antiviral neutralization of sotrovimab against the BA.2 subvariant.
  Other Names: VIR-7831

SUMMARY:
This is an open-label study examining the safety and tolerability of sotrovimab, administered in two sequential doses as prophylaxis in immunocompromised patients with impaired humoral immunity against SARS-CoV-2.

DETAILED DESCRIPTION:
This open-label study evaluated the safety and tolerability of sotrovimab, administered in two sequential doses, as COVID-19 prophylaxis in immunocompromised patients with impaired humoral immunity against SARS-CoV-2. 93 patients were enrolled in this study, 10 patients in an initial lead-in PK cohort initially planned to determine the optimal dosing interval between the first and second dose of sotrovimab and assess the safety and tolerability of the drug (prior to the spread of the BA.2 variant, which made it necessary to administer the repeat sotrovimab dose earlier than originally anticipated, using theoretical modeling and logistical considerations), 50 patients (including the 10 patients in the lead-in PK cohort) in a safety and tolerability lead-in cohort to examine rates of infusion-related reactions (IRR) with a 30-minute sotrovimab IV infusion, and the remainder in an expansion cohort for further assessment of the safety and tolerability of sotrovimab in this patient population, with the sotrovimab infusion duration determined by the rate of IRRs in the 50-patient safety and tolerability lead-in cohort. The first treatment consisted of sotrovimab 500mg as an intravenous (IV) infusion over 30 minutes, followed by a one-hour monitoring period. The second treatment, administered in a time when BA.2 became the dominant SARS-CoV-2 variant, consisted of sotrovimab 2000mg as an intravenous (IV) infusion over 60 minutes, followed by a two-hour monitoring period in the first 10 patients administered this dose, who comprised a second lead-in safety cohort for this 2000mg dose, and a one-hour monitoring period in all patients subsequently receiving their second sotrovimab dose, maintaining this one-hour monitoring period as long as there were no grade >2 infusion-related reactions or other SAEs potentially related to the sotrovimab dose in this 2000mg dose lead-in safety cohort.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age or older at the time of consent and weigh at least 40 kg. Children will be excluded from this study because dosing and adverse event data are limited for the use of sotrovimab in participants <18 years of age.
* Participant must have one of the following immunocompromising conditions that increases their likelihood of having an impaired humoral immune response to SARS-CoV-2, while also increasing their risk of being infected with SARS-CoV-2 and risk of progression to severe COVID-19:

  1. Exposure to an anti-CD20 monoclonal antibody (e.g. all formulations of rituximab, obinutuzumab, ofatumumab, ocrelizumab, ibritumomab, tositumomab) for a hematologic malignancy or an autoimmune/inflammatory disease in the 12-month period prior to consent.
  2. Allogeneic hematopoietic cell transplant ≥ 3 months and ≤ 1 year prior to consent; or allogeneic hematopoietic cell transplant >1 year prior to consent plus active graft-versus host disease on systemic immunosuppressive therapy.
  3. Chimeric antigen receptor (CAR)-T cell therapy ≥ 4 weeks and ≤ 2 years prior to consent.
  4. Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), multiple myeloma, or Waldenström macroglobulinemia.
  5. Solid organ transplant recipient receiving immunosuppressive therapy.
  6. Congenital immunodeficiency syndrome (e.g. Wiskott-Aldrich syndrome, DiGeorge syndrome, common variable immunodeficiency).
  7. Patients with hematologic malignancy or autoimmune/inflammatory disease exposed to immunosuppressive medications specifically associated with a blunted humoral immune response to SARS-CoV-2 vaccination (e.g. mycophenolate mofetil, azathioprine, methotrexate, Bruton tyrosine kinase inhibitors, ruxolitinib, venetoclax, or corticosteroids (prednisone >20mg or equivalent daily for at least 14 days) in the 3-month period prior to consent.
* Female participants must be:

  1. Postmenopausal for at least 1 year;
  2. Post-hysterectomy and/or post-bilateral oophorectomy;
  3. Of childbearing potential, with a negative urine or serum human chorionic gonadotropin pregnancy test prior to each sotrovimab dose, and agree to use a highly effective method of birth control throughout the study period.
* Participants must have a negative or low-positive (<50 U/mL) SARS-CoV-2 spike antibody assay result within 28 days of consent.

Exclusion Criteria:

* Participants with an active SARS-CoV-2 infection, with a positive SARS-CoV-2 RT-PCR or antigen test result within 21 days prior to consent.
* Participants with symptoms suggestive of SARS-CoV-2 infection.
* Close contact (less than 6 feet away for a cumulative total of ≥ 15 minutes over a 24-hour period) with an individual with COVID-19 in the 14 days prior to consent.
* Individuals who are pregnant or breastfeeding.
* Participants who are receiving any other investigational agents.
* Participants who, in the judgment of the investigator, are likely to have a life expectancy of less than one year.
* Known hypersensitivity to any constituent present in sotrovimab or any other anti-SARSCoV-2 monoclonal antibody product.
* Active enrollment on another interventional research study of any agent for the treatment or prophylaxis of SARS-CoV-2 infection.
* Exposure to any other anti-SARS-CoV-2 monoclonal antibody product for the treatment of COVID-19 in the prior 6 months.
* Exposure to any other anti-SARS-CoV-2 monoclonal antibody product for prophylaxis against COVID-19 infection in the prior 12 months.
* Receipt of a SARS-CoV-2 vaccine dose within the prior 28 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Koo, MD, Principal Investigator — Dana-Farber/Brigham and Women's Cancer Center; Jennifer Manne-Goehler, MD, ScD, Principal Investigator — Brigham and Women's Hospital; Sarah P Hammond, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Bocco IH, Beluch K, Cho A, Lahoud C, Reyes FA, Moshovitis DG, Unger-Mochrie GM, Wang W, Hammond SP, Manne-Goehler J, Koo S. Safety and tolerability study of sotrovimab (VIR-7831) prophylaxis against COVID-19 infection in immunocompromised individuals with impaired SARS-CoV-2 humoral immunity. Pilot Feasibility Stud. 2023 Jun 16;9(1):100. doi: 10.1186/s40814-023-01325-y. PMID 37328890

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no significant events in the study occurring after enrollment and prior to assignment into a group - this was a single arm safety and tolerability study.
Groups:
- Sotrovimab: Two intravenous (IV) doses of sotrovimab were administered in total - the first on Treatment Day 1 (500mg) and the second on Treatment Day 2, approximately 8-14 weeks after the first dose, at a higher 2000mg dose, in light of the reduced antiviral susceptibility of the BA.2 subvariant to sotrovimab, with the dosing interval determined by theoretical modeling of the duration of efficacy of sotrovimab as antiviral prophylaxis based on the rising prevalence of the Omicron BA.2 subvariant.
Period: Overall Study
Arm/Group | Sotrovimab
Started | 93
Completed | 88
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Sotrovimab
Number analyzed (Participants) | 93
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.4 [32.3 to 93.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 85
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 85
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 93

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Treatment-emergent Adverse Events, Serious Adverse Events, and Adverse Events of Specific Interest
Description: Proportion of patients with treatment-emergent adverse events, serious adverse events, and adverse events of specific interest (including infusion-related and hypersensitivity reactions, anti-drug antibody (ADA) levels, and antibody-dependent enhancement
Time Frame: 36 weeks after the second dose of sotrovimab
Population: immunocompromised patients with impaired humoral immunity to SARS-CoV-2
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab
Number analyzed (Participants) | 93
Participants
  Proportion of subjects with treatment-emergent grade 3-4 adverse events, per DAIDS grading criteria. | 28
  Proportion of study subjects with treatment-emergent serious adverse events (SAE). | 27
  Proportion of study subjects with infusion-related and hypersensitivity reactions | 3
  Proportion of study subjects with the development of antidrug antibody (ADA) levels | 3
  Proportion of subjects with antibody-dependent enhancement (ADE) | 0

2. Primary Outcome: Half-life of Sotrovimab in Immunocompromised Patients With Impaired Humoral Immunity Against SARS-CoV-2.
Description: Evaluation of half-life of sotrovimab in immunocompromised patients with impaired humoral immunity against SARS-CoV-2.
Time Frame: Within 1 hour of the first dose infusion of sotrovimab and on day 11, 29, and 59. Prior to the second dose, within 1 hour of the second dose infusion of sotrovimab, and 11, 29, 59, and 168 days after
Population: immunocompromised patients with impaired humoral immunity against SARS-CoV-2, range reported is a 5-95th percentile
Measure: Median (90% Confidence Interval); unit: days (half-life)
Arm/Group | Sotrovimab
Number analyzed (Participants) | 93
days (half-life) | 67.7 [47.3 to 95.8]

3. Secondary Outcome: COVID-19-related Outcomes
Description: The proportion of study subjects who: (a) develop COVID-19 (of any severity), (b) severe COVID-19, (c) Emergency department (ED) visits, inpatient hospitalization, or ICU hospitalizations within 28 days of a new diagnosis of SARS-CoV-2, (d) need for new or increasing supplemental oxygen or mechanical ventilation within 28 days of a new diagnosis of SARS-CoV-2, and (e) death due to any cause during the study follow-up period.
Time Frame: 36 weeks after the second dose of sotrovimab
Population: immunocompromised patients with an impaired humoral immune response to SARS-CoV-2
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab
Number analyzed (Participants) | 93
Participants
  Patients who developed COVID-19 (of any severity) | 35
  Patients who developed severe COVID-19 | 1

4. Secondary Outcome: General Health Quality of Life Measurement
Description: Health-related quality of life was assessed using the 36-Item Short Form Survey (SF-36), specifically focusing on the General Health domain. Each question in this domain was scored as follows:
  For questions 33 and 35, responses were scaled: 1 = 0, 2 = 25, 3 = 50, 4 = 75, and 5 = 100.
  For questions 1, 34, and 36, responses were scaled: 1 = 100, 2 = 75, 3 = 50, 4 = 25, and 5 = 0.
  The scores for these five questions were summed to create a composite General Health score, with possible total scores ranging from 0 (indicating the best perceived general health) to 500 (indicating the worst perceived general health). Lower scores indicate better perceived general health.
  We calculated the mean General Health score at two time points: treatment day 1 and treatment day 2. The reported results reflect the difference between these mean scores, with negative differences indicating improvement and positive differences indicating a decline in p
Time Frame: At treatment day 1, at treatment day 2
Population: immunocompromised patients with impaired humoral immunity to SARS-CoV-2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sotrovimab
Number analyzed (Participants) | 93
scores on a scale | -0.60 (3.27)

5. Secondary Outcome: In Patients Who Develop COVID-19, the Greatest Extent of COVID-19 Symptoms, as Assessed Using the 8-point National Institute of Allergy and Infectious Diseases Ordinal Scale (NIAID-OS)
Description: National Institute of Allergy and Infectious Disease Ordinal Scale (NIAD-OS) was assessed at the end of hospitalization or 14 days after the diagnosis of COVID-19. The worst reported scale value was used in the analysis to adequately represent the greatest extent of their COVID-19 infection.
  NIAID-OS Scale Value Description
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities or/or requiring home oxygen
  3. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care
  4. Hospitalized, not requiring supplemental oxygen
  5. Hospitalized, requiring supplemental oxygen
  6. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  7. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  8. Death
Time Frame: from covid day 1 to end of hospitalization or covid day 14
Population: study subjects who acquired SARS-CoV-2 during the study period
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Sotrovimab
Number analyzed (Participants) | 35
units on a scale | 1 [1 to 5]

6. Other Pre Specified Outcome: Number of Participants With New Cellular or Antibody-mediated Rejection Events
Description: Assessment of rates of new cellular or antibody-mediated rejection events in solid organ transplant (SOT) recipients exposed to sotrovimab.
Time Frame: 36 weeks after the second dose of sotrovimab
Population: immunocompromised patients with impaired humoral immunity to SARS-CoV-2
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab
Number analyzed (Participants) | 93
Participants | 0

7. Other Pre Specified Outcome: New-onset or Worsening Graft-versus-host Disease in Hematopoietic Cell Transplant Recipients
Description: Assessment of rates of new-onset or worsening graft-versus-host disease in hematopoietic cell transplant (HCT) recipients exposed to sotrovimab.
Time Frame: 36 weeks after the second dose of sotrovimab
Population: immunocompromised patients with impaired humoral immunity to SARS-CoV-2
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab
Number analyzed (Participants) | 93
Participants | 0

8. Other Pre Specified Outcome: New-onset Allograft or Stem Cell Failure Requiring Retransplantation in HCT Recipients
Description: Assessment of rates of new-onset allograft or stem cell failure requiring retransplantation in HCT recipients exposed to sotrovimab.
Time Frame: 36 weeks after the second dose of sotrovimab
Population: immunocompromised patients with impaired humoral immunity to SARS-CoV-2
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab
Number analyzed (Participants) | 93
Participants | 0

ADVERSE EVENTS:
Time Frame: 68-74 weeks
Description: Study subjects were assessed according to the study calendar in the protocol: regular laboratory testing, scheduled investigator assessments, and scheduled questionnaires.
Groups:
- Sotrovimab: Two intravenous (IV) doses of sotrovimab were be administered in total - the first on Treatment Day 1 (500mg) and the second on Treatment Day 2, approximately 8-14 weeks after the first dose, at a higher 2000mg dose, in light of the reduced antiviral susceptibility of the BA.2 subvariant to sotrovimab, with the dosing interval determined by theoretical modeling of the duration of efficacy of sotrovimab as antiviral prophylaxis based on the rising prevalence of the Omicron BA.2 subvariant.
  Sotrovimab: Two intravenous (IV) doses of sotrovimab were administered over the study period, the first 500mg, and the second 2000mg, in light of the reduced antiviral neutralization of sotrovimab against the BA.2 subvariant, which became the dominant variant in between the administration of the two doses.
Arm/Group | Sotrovimab
All-Cause Mortality (participants affected / at risk) | 1/93
Serious Adverse Events (participants affected / at risk) | 27/93
Other Adverse Events (participants affected / at risk) | 10/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sotrovimab (N=93)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Heart Failure (Cardiac disorders) | 2
Non-St Elevation Myocardial Infarction (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Upper GI Bleed (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Empyema (Infections and infestations) | 1
COVID-19 infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Tracheobronchitis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 1
Worsening Pneumonia (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Burn Scar In The Bronchus (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sotrovimab (N=93)
Pneumonia (Infections and infestations) | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT05210101/Prot_SAP_000.pdf